CLINICAL TRIAL: NCT02643095
Title: Efficacy of Scleral Contact Lenses for Daily Wear for Regular and Irregular Refractive Errors Compared to Habitually Worn Scleral Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Fogt (Other)
Responsible Party: Sponsor-Investigator, Jennifer Fogt, Assistant Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015W0197
Record Dates: First submitted 2015-12-28; First posted 2015-12-30 (Estimated); Results first posted 2018-09-13 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Scleral Lens Wearers

ARMS (1):
- Lens fitting/evaluation (Experimental): This study will be done with subjects who already habitually wear scleral contact lenses. The study lens is made with a material that is already widely available and has a new design. It will be fit by the investigators and will be assessed and at one week and 1 month.
  Interventions: Device: scleral contact lens

INTERVENTIONS:
Device: scleral contact lens — Scleral contact lens

SUMMARY:
This study will be done with subjects who already habitually wear scleral contact lenses. The study lens is made with a material that is already widely available and has a new design. It will be fit by the investigators and will be assessed and at one week and 1 month.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects may be male or female, of any race, and at least 18 years old at the time of the pre-treatment examination.
2. Subjects must habitually wear scleral contact lenses for an average wearing time of 6 hours per day.
3. The prospective eye(s) must have refractive hyperopia or myopia from +20.00 to -20.00 diopters sphere (spectacle plane), with up to -10.00 diopters of refractive astigmatism (spectacle plane), as determined by manifest refraction (phoropter or trial frame with a 12.5 mm vertex distance).
4. Subjects must have best spectacle corrected visual acuity of at least 0.5 logMAR in each eye.
5. Subjects must be willing and capable to return for all scheduled follow-up visits for a period of at least 3 months (minimum of 1 month from initial dispensing).

Exclusion Criteria:

1. Female subjects who are pregnant, breast-feeding or intend to become pregnant over the course of the study.
2. Subjects with a history of any of the following medical conditions: collagen vascular disease, autoimmune disease, immunodeficiency diseases, ocular herpes zoster or simplex, endocrine disorders (including, but not limited to active thyroid disorders and diabetes), lupus, and rheumatoid arthritis.

   Note: The presence of diabetes (either type 1 or 2), regardless of disease duration, severity or control, will specifically exclude subjects from eligibility.
3. Subjects with active ophthalmic disease or abnormality including glaucoma, chorioretinitis, central retinal artery or vein occlusion, intraocular or ocular infection.
4. Subjects who are participating in any other clinical trial (FDA or other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-01-26 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-08-31 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens Fitting/Evaluation: This study was conducted with subjects who already habitually wore scleral contact lenses. The study lens was made with a material that is already widely available and has a new design. It was fit by the investigators and assessed one week and 1 month of wear.
  scleral contact lens: Scleral contact lens
Period: Overall Study
Arm/Group | Lens Fitting/Evaluation
Started | 22
Completed | 21
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Lens Fitting/Evaluation: This study was conducted with subjects who already habitually wear scleral contact lenses. The study lens is made with a material that is already widely available and has a new design. It was fit by the investigators and assessed and at one week and 1 month.
  scleral contact lens: Scleral contact lens
Arm/Group | Lens Fitting/Evaluation
Number analyzed (Participants) | 22
Age, Customized [Count of Participants; unit: Participants]
  Age 18 or older | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint of the Study is the Overall Satisfaction and Desire to Continue Wearing the Study Lenses
Description: Number of Participants with Overall Satisfaction and Desire to Continue Wearing the Study Lenses
Time Frame: 1 month after lens is dispensed
Measure: Count of Participants; unit: Participants
Arm/Group | Lens Fitting/Evaluation
Number analyzed (Participants) | 21
Participants
  Preferred test lenses to habitual lenses | 15
  Preferred habitual lenses to test lenses | 2
  No preference | 4

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at all study visits, including a visit after 1 week and 1 month of lens wear.
Arm/Group | Lens Fitting/Evaluation
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 1/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens Fitting/Evaluation (N=21)
punctate keratitis (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No